CLINICAL TRIAL: NCT03716245
Title: A Multicenter, Randomised, Open-label Prospective Clinical Trial to Evaluate the Clinical Significance of Supraclavicular Lymph Node Dissection for Breast Cancer Patients With Ipsilateral Supraclavicular Lymph Node Metastasis
Brief Title: Clinical Significance of Supraclavicular Lymph Node Dissection for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhong Wu, PhD (Other)
Responsible Party: Sponsor-Investigator, Xinhong Wu, PhD, vice-president, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLND0919
Record Dates: First submitted 2018-10-14; First posted 2018-10-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Stage III
Keywords: breast cancer; supraclavicular lymph node; dissection; radiotherpy; prognosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supraclavicular lymph node dissection and raidiotherapy (Experimental): breast cancer patients with supraclavicular lymph node metastasis receive supraclavicular lymph node dissection and supraclavicular area radiotherapy
  Interventions: Procedure: supraclavicular lymph node dissection
- supraclavicular area radiotherapy (Active Comparator): breast cancer patients with supraclavicular lymph node metastasis receive supraclavicular area radiotherapy
  Interventions: Radiation: supraclavicular area radiotherapy

INTERVENTIONS:
Procedure: supraclavicular lymph node dissection — people with supraclavicular lymph node metastasis before surgery should receive dissection of supraclavicular lymph node and the supraclavicular lymph node metastasis should be confirmed either by core needle biopsy or fine needle aspiration biopsy
  Arms: supraclavicular lymph node dissection and raidiotherapy
Radiation: supraclavicular area radiotherapy — people with supraclavicular lymph node metastasis before surgery should receive radiotherapy of supraclavicular area and the supraclavicular lymph node metastasis should be confirmed either by core needle biopsy or fine needle aspiration biopsy
  Arms: supraclavicular area radiotherapy

SUMMARY:
Breast cancer patients with ipsilateral supraclavicular lymph node metastasis are defined as Ⅲc stage (N3) according to the newly published 8th AJCC TNM staging system. No concret guide line was supported to such patients. It is still pending whether to exert supraclavicular lymph node dissection to breast cancer patients with ipsilateral supraclavicular lymph node metastasis.

To evaluate the clinical significance and complication of supraclavicular lymph node dissection for breast cancer patients with ipsilateral supraclavicular lymph node metastasis, the investigators randomize patients into two groups, one group is supraclavicular lymph node dissection with radiotherapy group, the other group is radiotherapy group.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer and the leading cause of deaths from cancer in women worldwide. Breast cancer patients with ipsilateral supraclavicular lymph node metastasis are defined as Ⅲc stage (N3) according to the newly published 8th AJCC TNM staging system. Clinical outcomes are similar for patients with ipsilateral supraclavicular lymph node metastases at first presentation and for patients with recurrent ipsilateral supraclavicular lymph node metastases. The survival rate was lower in patients with ipsilateral supraclavicular lymph node metastases than in patients with lower axillary or subclavian nodal involvement. No concrete guide line was supported to such patients. It is still pending whether to exert supraclavicular lymph node dissection to breast cancer patients with ipsilateral supraclavicular lymph node metastasis. Patients with ipsilateral supraclavicular lymph node metastases who were treated with surgery or radiotherapy and achieved good neck control were reported to achieve better survival than those for whom surgical treatment or irradiation did not result in good local control.

Patients with ipsilateral supraclavicular lymph node metastases should be offered a combined modality approach, including systemic therapy, surgery, and radiotherapy. Furthermore, local treatment, usually including axillary and supraclavicular lymph node, either by surgical clearance or by radical radiotherapy, can prevent the tumor cells from drainage, might be play a more important role. However, the role of surgical removal of the supraclavicular nodes is uncertain compared with radical radiotherapy. To our knowledge, the available literature comparing these two local treatments of ipsilateral supraclavicular lymph node metastases is scarce. Furthermore, the studies comparing the outcome of dissection of supraclavicular lymph node combined with local radiotherapy and radiotherapy of supraclavicular lymph node is also rare. All the related reports up to date have mixed them up.

To evaluate the clinical significance and complication of supraclavicular lymph node dissection for breast cancer patients with ipsilateral supraclavicular lymph node metastasis, we randomize patients into two groups, one group is supraclavicular lymph node dissection with radiotherapy group, the other group is radiotherapy group.

Therefore, in addition to investigating the role of surgical removal of the supraclavicular nodes in Chinese patients, we also try to reveal the potential difference between these two treatments, hoping to bring more insight into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study procedures and contents, and willingness to voluntarily sign the written informed consent form;
2. Age≤75 years old, female;
3. Histologically confirmed breast cancer;
4. Histologically or cytologically confirmed ipsilateral supraclavicular lymph node metastasis；
5. cT0-T3；
6. low and moderate risk for anesthesia

Exclusion Criteria:

1. Absolute and relative contraindication for surgery or radiation；
2. existing distant metastasis before surgery；
3. non-invasive breast cancer；
4. with contralateral breast cancer；
5. Previous history of breast cancer or other malignancies；
6. ECOG≥2；
7. inflammatory breast cancer；
8. pregnancy；
9. any serious complications which caused patients not suitable to participate this study

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 180 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 3-5 years
  Disease free survival for 3 years and 5 years, which means the rate of patients without local recurrence and distant metastasis in the whole patients at the same group will be calculated with Kaplan Meier survival curves.

SECONDARY OUTCOMES:
Occurring rate of complications | 3-5 years
  Occurring rate of complications including the occurring rate of infection, hemorrhage, limb lymphedema, time in hospital, brachial plexopahy, radiation induced lung injury in each group were recorded in patients' medical record.
Overall survival | 3-5 years
  Overall survival for 3 years and 5 years, which means the rate of patients alive in the whole patients at the same group will be calculated with kaplan meier survival curves.
Life quality score | 3-5 years
  Life quality score was evaluated by European Organization of Research and treatment of Cancer-Questionnaire of Life Quality-C30 Version 3 (EORTC-QLQ-C30 V3), which conduct a series of questions about the patients' physical condition, activity of daily life, adverse reaction and mood condition. The range in the questionnaire for the score is from 1 to 4, in which 1 stands for having no discomfort and 4 stands for having great discomfort.
Recurrence free survival | 3-5 years
  Recurrence free survival for 3 years and 5 years, which means the rate of patients without local recurrence in the whole patients at the same group will be calculated with Kaplan Meier survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Xinhong Wu, Doctor, Principal Investigator — Hubei Cancer Hospital
Locations (1):
- Wu Xinhong, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code